CLINICAL TRIAL: NCT05871047
Title: Prevalence of Nerd Neck Between Different Students at Taibah University, Saudi Arabia; Cross Section Design
Brief Title: Prevalence of Nerd Neck Between Different Students at Taibah University, Saudi Arabia
Status: Completed | Type: Observational
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, walaa M Ragab, assistant professor, Taibah University
Other Study IDs: wragab
Record Dates: First submitted 2023-04-30; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: CERVICAL

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- practical group
  Interventions: Device: tragus to wall distance (TWD), craniovertebral angle (CVA) by smart phone application
- non-practical group
  Interventions: Device: tragus to wall distance (TWD), craniovertebral angle (CVA) by smart phone application

INTERVENTIONS:
Device: tragus to wall distance (TWD), craniovertebral angle (CVA) by smart phone application — Applying photogrammetric method for CVA by smart phone application and measure nerd neck objectively from both sitting and standing positions. Also, tragus to wall distance method was used to detect degree of nerd neck from the standing position.

SUMMARY:
A convenient sample of 82 female students aged 18-24 years participated in analytic observational experiment cross section design. Students were recruited into two groups, practical and non-practical. to answer the following

1. Is there a difference in the prevalence of nerd neck between students of practical and non-practical studying groups at Taibah University from the sitting position?
2. Is there a difference in the prevalence of nerd neck between students of practical and non-practical studying groups at Taibah University from the standing position?

ELIGIBILITY:
Inclusion Criteria:

* A convenient sample of 82 female students
* the age was between 18-24 years
* Students were recruited from practical and non-practical faculties at taibah university.

Exclusion Criteria:

* we excluded Any student with previous neck or back surgery or history of previous accident
* Also, any student with history of cervical column fracture injury, scoliosis, severe thoracic kyphosis, torticollis, persistent respiratory problems, rheumatic disease.
* also we excluded any student with loss of standing balance and user of hearing aid

Ages: 18 Years to 24 Years | Sex: Female
Age Groups: Adult
Study Population: Practical group was recruited from college of Medical Rehabilitation Sciences and Applied Medical Sciences while non-practical group was recruited from Business Administration. Posters, word of mouth, and WhatsApp groups were used to recruit both groups.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
the prevalence of nerd neck | one day
  we measured nerd neck by calculating CVA by tragus wall distance test from standing position

CONTACTS AND LOCATIONS:
Overall Officials: walaa M ragab, Principal Investigator — Taibah University
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No